CLINICAL TRIAL: NCT03957200
Title: Assessing Gestational Age in First Trimester Pregnancies: A Comparison of a New Handheld Wireless Transabdominal Ultrasound to a Portable Transabdominal Ultrasound
Brief Title: Assessing Gestational Age in First Trimester Pregnancies Using Ultrasound
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Helen Pymar, Associate Professor, University of Manitoba
Other Study IDs: HS22818 (B2019:034)
Record Dates: First submitted 2019-05-13; First posted 2019-05-21 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Early
Keywords: Ultrasound; pregnancy; first trimester; dating

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to assess equivalency of the transabdominal Clarius handheld wifi C3 ultrasound (which uses Bluetooth to locate the ipad Mini 5 and then uses wifi direct to show the images) to the current standard of care in Women's Hospital outpatient department the portable Zonare ZS3 in patients presenting in the first trimester of pregnancy.

DETAILED DESCRIPTION:
This is a prospective study in which first trimester participants who are presenting to discuss termination of pregnancy, will consent to have an additional transabdominal ultrasound with the Clarius C3 immediately prior to their standard ultrasound which is performed to date their pregnancy. Participants who are presenting for medical abortion have been prescreened to be estimated to be less than 9 weeks GA. Participants who are being seen prior to surgical abortion will have been screened by nurses based on their last menstrual period or estimated time of conception to estimate their gestational age. Potential participants estimated to be less than 13 weeks GA, will be approached to see if they are interested in participating in the study before they are seen by their health care provider. The name, date of approach, and reason for decline of potential participants who refuse to participate will be documented. If agreeable, the participant will complete consent with a study nurse or medical student for the additional ultrasound.

Participants will then receive the 2 ultrasounds by the same health care provider with the Clarius C3 ultrasound first, then the standard care ultrasound. Occasionally, there may be a different provider doing the Clarius C3 ultrasound when the patient consents.

Participants will receive standard care for medical or surgical abortion. The following information will be documented from their chart:

Height and weight, age, Obstetrical history (Gravida, para, number cesareans, ectopic pregnancies, spontaneous abortions, therapeutic abortions). If they do not have a documented intrauterine pregnancy, the standard questions to rule out possibility of ectopic pregnancy will be determined, and any positive answers will be documented in the chart. Anyone without a documented intrauterine pregnancy (no gestational sac or a gestational sac with no definite crown rump length or yolk sac) will be followed until a final outcome is determined or they are lost to follow up. When the patient has a pregnancy of unknown location (no evidence of a pregnancy inside or outside of the uterus), their data will not be used to compare the two ultrasounds but future outcome will be recorded.

The final outcome of their pregnancy and any complications will be determined within the next 6 weeks with the following potential outcomes:

completed medical abortion, completed surgical abortion (possibily following failed medical abortion), lost to follow up, continuing pregnancy, or ectopic pregnancy.

If a participant is determined to be over 13 weeks GA, they will receive a dating ultrasound with the Clarius C3 ultrasound using biparietal diameter as appropriate but it will not be included in the final study measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting requesting medical or surgical abortion
2. Estimated to be under 13 weeks gestational age based on last menstrual period or time of conception, or nurses best estimate.
3. Able to provide informed consent with adult supervision of a minor or with an interpreter present

Exclusion Criteria:

1. Unable to provide informed consent

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients are presenting for an ultrasound prior to first trimester termination of pregnancy.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Womens Hospital- 735 Notre Dame Ave, Winnipeg, Manitoba
  - Women's Hospital 820 Sherbrook St (moved hospitals Dec 2019), Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van den Hof MC, Smithies M, Nevo O, Oullet A. No. 375-Clinical Practice Guideline on the Use of First Trimester Ultrasound. J Obstet Gynaecol Can. 2019 Mar;41(3):388-395. doi: 10.1016/j.jogc.2018.09.020. PMID 30784569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 patients were approached and 57 were eligible and provided consent.
Groups:
- Patients Received Ultrasound With Clarius Followed by Ultrasound With Zonare: Transabdominal ultrasound performed with Clarius handheld ultrasound followed by portable ultrasound Zonare ZS3
Period: Overall Study
Arm/Group | Patients Received Ultrasound With Clarius Followed by Ultrasound With Zonare
Started | 57
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 57 patients consented but information study information was reviewed when they were not Pregnancy of Unknown Location or over 13 weeks' gestational age (51)
Arm/Group | Patients Received Ultrasound With Clarius Followed by Ultrasound With Zonare
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only included those with no pregnancy of unknown location or gestational age under 13 weeks GA
  years
    number analyzed (Participants) | 51
    (all) | 29.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Can Both Transabdominal Ultrasounds See a Gestational Sac and Yolk Sac or Embryo?
Description: Number of participants with both ultrasounds showing a gestational sac with a yolk sac or embryo
Time Frame: Results will be known immediately after both ultrasounds are completed
Measure: Count of Participants; unit: Participants
Groups:
- Both Definite IUP, Both SAC Seen, Zonare Saw Definite IUP Where Clarius Saw Sac: Women under 13 weeks of gestational age.
Arm/Group | Both Definite IUP, Both SAC Seen, Zonare Saw Definite IUP Where Clarius Saw Sac
Number analyzed (Participants) | 51
Participants | 51

2. Secondary Outcome: Can Both Transabdominal Ultrasounds Give a Crown Rump Length or Gestational Sac Size to Within 5 Days
Description: Number of participants with both ultrasounds showing a crown rump length or gestational sac measurement within 5 days of error.
Time Frame: Results will be known immediately after both are completed
Reporting Status: Not Posted, anticipated posting 2025-07

ADVERSE EVENTS:
Time Frame: 36 weeks
Description: No concerns for adverse events related to participating
Arm/Group | Patients Received Ultrasound With Clarius Followed by Ultrasound With Zonare
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT03957200/Prot_SAP_000.pdf